CLINICAL TRIAL: NCT04021849
Title: Evaluation of a Virtual Course to Increase Knowledge in Sexual Harassment, Prevention and Sanction Policies of Cayetano Heredia Peruvian University in Pupils of the Faculty of Public Health and Administration: a Randomized Controlled Trial
Brief Title: Evaluation of Virtual Course to Increase Knowledge in Sexual Harassment,Prevention and Sanction Policies of a University
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Mireya Reyna Martínez Ipanaqué, Principal Investigator, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 103921
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Sexual Harassment
Keywords: Sexual Harassment; Virtual Course; Training
MeSH Terms: conditions — Sexual Harassment

STUDY DESIGN:
Intervention Model Description: Students will be randomly assigned to one of two groups until a total of 134 participants are recruited: 67 in the intervention group and 67 in the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be gathered in a classroom with computers to receive an asynchronous virtual class of 45 minutes, 1 pre-test, 1 post-test and satisfaction surveys with Likert scale. This session will take 2 hours approximately. After a month, they will take a second post-test to measure retention of knowledge. The pre-test and post-tests are all the same and they all will be taken by using computer.
  Interventions: Other: Asynchronous Virtual Class
- Control (Sham Comparator): Participants will be gathered in a classroom with computers to receive a face-to-face class of 45 minutes, 1 pre-test, 1 post-test and satisfaction surveys with Likert scale. This session will take 2 hours approximately. After a month, they will take a second post-test to measure retention of knowledge. The pre-test and post-tests are all the same and they all will be taken by using computer.
  Interventions: Other: Face-to-face Class

INTERVENTIONS:
Other: Face-to-face Class — The principal investigator will dictate a course about Sexual Harassment, Prevention and Sanction Policies of Cayetano Heredia Peruvian University using PowerPoint Presentation
  Arms: Control
Other: Asynchronous Virtual Class — Every student will have the access to a platform with an Asynchronous Virtual Class that will use the same PowerPoint Presentation of the intervention with an audio recorded by the principal investigator
  Arms: Intervention

SUMMARY:
Sexual harassment is the behavior of sexual or sexist connotation unwanted by the affected person. Despite being considered as gender-based violence, victims of sexual harassment can be of both sexes. The university is the most frequent place where university students suffer sexual harassment. Law No. 27942 - "Ley de Prevención y Sanción del Hostigamiento Sexual" and its amendments, includes training and prevention in sexual harassment. The Universidad Peruana Cayetano Heredia (UPCH) has a regulation for the prevention and punishment of sexual harassment. Education through the use of Information and Communications Technologies (ICT) is presented as an alternative to face-to-face classes, optimizing resources and achieving greater scope. The early, mandatory and massive dissemination at the university of a training in sexual harassment could be achieved through a virtual course. However, there is little research on the evaluation of the effectiveness of prevention programs in sexual violence in university students. The objective is to prove that taking a virtual course about sexual harassment, prevention and sanction policies of the UPCH can achieve a greater or same knowledge of the subject in the students of the UPCH, compared to a face-to-face course. The study design is a randomized controlled trial to assess the level of knowledge in this subject, whose control group is provided classes in face-to-face mode. Also, both modalities of the course will include a survey with Likert scale to measure the degree of satisfaction with the course taken. And finally, it includes a qualitative study through focus groups with the university students of the classroom and virtual classes to know their appreciations of both modalities of the course.

DETAILED DESCRIPTION:
Main Objective:

Compare the improvement of knowledge about sexual harassment, prevention and sanction policies of the UPCH of the asynchronous virtual course with the face-to-face course in students of the UPCH.

Study Design:

A randomized control trial will compare the improvement of knowledge among who received asynchronous virtual classes and those who received face-to-face classes by applying a pre-test and 2 post-test. The pre-test and the first post-test will be taken the day of the intervention and the second post-test will be taken after a month to measure knowledge retention.

To measure the degree of satisfaction with the course modality, the intervention's day the students will take a survey with Likert scale. And separately, some students of the intervention and control group will be interview in focus groups to know their appreciations about the satisfaction perceived with the modality of the course taken.

Population:

Undergraduate university students enrolled in the 2019-II period of the Faculty of Public Health and Administration (FASPA).

Sample:

For the randomized control trial, a sample of 67 participants per group was calculated with a significance of 95%, a power of 80% and a loss of follow-up rate of 6%, to show a difference of 7% in the scores of knowledge of sexual harassment between the two groups.

For the qualitative analysis of the focus groups, for each course modality, there will be two sessions of 6 people who completed the course. However, focus groups will continue to be carried out until the sample becomes saturated, that is, until the information obtained from these meetings is redundant or the objectives of the study are clarified.

Group assignment:

Students of FASPA will be invited to participate by flyers and invitations in classrooms. Also, by e-mail they will receive an invitation with the informational consent form and a link to fill out a registration form for the ones who are interested in participating. If inclusion and exclusion criteria are met, students will be accepted to participate in the study and they will be randomly assigned to one of the two groups. Finally they will receive an e-mail confirming their participation and the available schedules for the classes.

Ethical considerations:

Students who are registered and want to participate but do not meet the inclusion and exclusion criteria of the study, will be offered the virtual course restricting the access to the evaluations.

Every participant will receive the informational consent form. Data confidentiality will be maintained. Personal identifiers will be stored in a separate database, which will be password protected and accessible only to the research team. At the end of this project, UPCH will be able to dispose of the virtual course developed in this study for the purposes that may be appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate university students enrolled in the 2019-II period of FASPA

Exclusion Criteria:

* Students who have already taken a course on sexual harassment
* Exchange students (foreigners)
* Students who have not completed the pre-test and post-tests

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Level of Knowledge about sexual harassment | 3 months
  Measured by the automatic score the student get after taking the tests in a web platform.
  The instrument is a questionnaire made up of 20 multiple-choice questions about knowledge in sexual harassment, prevention and sanction policies of the university. Each correct question is worth 5 points so the scale range will be 0-100 points in total but then it will be converted to vigesimal score from 0 to 20 points, being the passing grade 11.00.

SECONDARY OUTCOMES:
Satisfaction with the course measured by a Likert-scale survey | 3 months
  Number of positive responses / total number of questions. The instrument is a Likert-scale survey with 9 questions about how satisfied is the student with the class session, the trainer, the class duration, the web platform, the quality of the class and others. The possible answers are: "Nothing", "Something", "A lot" and "Totally". Being the positive responses "A lot" and "Totally".
Satisfaction with the course described by a qualitative analysis of focal groups | 3 months
  The focal groups will be carried out with the students of the 2 course modalities, separately. The instrument for this focus group is a questionnaire about the satisfaction with the modality of the course, the content of the course and the fulfillment of expectations of the students on the course, the trainer and the web platform.

CONTACTS AND LOCATIONS:
Overall Officials: Mireya R Martínez Ipanaqué, B.E., Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (1):
- Universidad Peruana Cayetano Heredia, San Martín de Porres, Lima region, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zapp D, Buelow R, Soutiea L, Berkowitz A, DeJong W. Exploring the Potential Campus-Level Impact of Online Universal Sexual Assault Prevention Education. J Interpers Violence. 2021 Mar;36(5-6):NP2324-NP2345. doi: 10.1177/0886260518762449. Epub 2018 Mar 26. PMID 29577841
- [Background] Banyard VL, Moynihan MM, Plante EG. Sexual violence prevention through bystander education: an experimental evaluation. J Community Psychol [Internet]. 2007 [cited 2019 Feb 20];35(4):463-481. Available from: http://www.ncdsv.org/images/Sex%20Violence%20Prevention%20through%20Bystander%20Education.pdf
- [Background] Ley de Prevención y Sanción del Hostigamiento Sexual. Ley N° 27942. Publicado en el diario oficial El Peruano, (05 de Febrero de 2003).
- [Background] Decreto legislativo que incorpora el delito de acoso, acoso sexual, chantaje sexual y difusión de imágenes, materiales audiovisuales o audios con contenido sexual al código penal, y modifica el procedimiento de sanción del hostigamiento sexual. Decreto Legislativo N° 1410. Publicado en el diario oficial El Peruano, (11 de Septiembre de 2018).
- [Background] Bardales O, Ortiz Z. Hostigamiento sexual en mujeres y varones universitarios. Estudio exploratorio [Internet]. Lima: MIMP;2012 [cited 2019 Jan 14]. Available from: http://redin.pncvfs.gob.pe/images/publicacion2/hostigamiento-sexual-en-mujeres-y-varones-universitarios9.pdf
- [Background] Sarmiento P, Marcelo Y, Revollar E. Aproximación a la problemática del hostigamiento sexual laboral contra mujeres. Supervisión a ministerios, gobiernos regionales y Poder Judicial [Internet]. Lima: Defensoría del Pueblo del Perú; 2018 [cited 2019 Jan 14] Serie Informe de Adjuntía - Informe N° 007 - 2018- DP/ADM. Available from: https://www.defensoria.gob.pe/wp-content/uploads/2018/07/Informe-de-Adjuntia-007-2018-DP-ADM-II.pdf
- [Background] Loli S. La Prevención y Sanción del Hostigamiento Sexual. Módulo de asistencia técnica para el abordaje desde la perspectiva de género [Internet]. Lima: MIMDES; 2008 [cited 2019 Jan 20]. Available from: https://www.mimp.gob.pe/files/direcciones/dgignd/publicaciones/prevencion_sancion_hostigamiento_sexual_modulo_ACDI.pdf
- [Background] Carvajal Z, Delvó P. Análisis comparativo de dos estudios sobre hostigamiento sexual en la población estudiantil de la universidad nacional. Rev Latinoam Derechos Humanos [Internet]. 2010 [cited 2019 Jan 22];21(2):83-104. Available from: http://www.revistas.una.ac.cr/index.php/derechoshumanos/article/view/1930/1832
- [Background] Ministerio de Trabajo y Promoción del Empleo. Guía para prevenir el hostigamiento sexual en el ámbito laboral [Internet]. Lima: MTPE; 2011[cited 2019 Jan 20]. Available from: http://www.academia.edu/13809973/Ministerio_de_Trabajo_y_Promoción_del_Empleo